CLINICAL TRIAL: NCT05656378
Title: A Repository to Study Host-Microbiome Interactions in Health and Disease
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10001146; 001146-I
Record Dates: First submitted 2022-12-15; First posted 2022-12-19 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-10-01

CONDITIONS: Healthy Controls; Pregnancy; Pediatric Illnesses; Inflammatory Diseases
Keywords: Microbiome; Host Response; Children; Pregnancy; Natural History

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single Cohort: Participants aged >0 years with no upper age limit, both healthy volunteers and those with previously known and unknown disease states

SUMMARY:
Background:

The microbiome is the bacteria and other microorganisms that live inside and on the body. The microbiome is important for our health. Researchers study how the microbiome help people stay healthy. They study how the microbiome affects the body when people get sick. To do this research, they need samples of the microbiome living on the bodies of many people. The purpose of this natural history study is to collect microbiome samples in a repository. These samples will be used for future research.

Objective:

To collect microbiome samples from the body that can be used for future research.

Eligibility:

People of any age. Only those older than 3 years will be seen at the NIH clinic.

Design:

Participants will fill out a questionnaire. Topics will include their medical history and foods they eat.

Participants will be asked to give 1 or more of the following:

Stool, urine, saliva, vaginal fluid, and breastmilk. These samples can be collected at home and sent to the researchers.

Cells from participants cheek, nose, mouth, skin, rectum, and/or vagina. The cells may be collected by rubbing the area with a sterile cotton swab. These procedures can also be done at home.

Blood. Blood may be drawn using a needle inserted into a vein in the arm. For young children, blood may be collected by a prick on the heel or finger.

Intestinal tissue samples. These may be collected from participants who are having an endoscopy or colonoscopy for other reasons.

Skin tissue samples. These may be collected from participants who are having biopsies for other reasons.

...

DETAILED DESCRIPTION:
Study Description:

The human microbiome and host response to the microbiome play a key role in human health and disease. The Clinical Microbiome Unit focuses on clinical microbiome intervention trials to improve human health. This is a sample collection repository protocol to provide samples needed for validation of assays and techniques vital to the success of designing and analyzing interventional trials.

Primary Objective:

To collect biological specimens to assess host microbiome response for 1) assay validation, 2) optimization of techniques for collection, storage, processing and analyzing samples, 3) control samples for research tests in other studies, and 4) identification of potential targets from which clinical trials can be designed to better understand or mitigate microbiome-associated diseases.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Aged >0 years. Only participants >3 years old will be seen at the NIH CC.
* Willing to allow biological samples and data to be stored for future research.
* Willing to provide at least one of the requested biospecimens.

EXCLUSION CRITERIA:

* An individual who has any condition that, in the judgment of the investigator, may put them at undue risk or make them unsuitable for participation in the study will be excluded.
* For additional gastrointestinal and skin biopsies only, individuals on blood thinners unless they have already been stopped for the procedure.
* For additional gastrointestinal biopsies only, individuals who have a history of gastrointestinal perforation with endoscopic biopsies will be excluded from the collection of additional gastrointestinal biopsies for the repository.
* For additional gastrointestinal biopsies only, healthy children (<18 years old).
* For skin biopsies only, individuals who have a history of keloid formation.
* For vaginal swabs and vaginal fluid only, individuals who have not started menses.
* For breast milk only, non-lactating individuals.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: People of all ages who meet study criteria.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-03-09 (Actual); Primary Completion 2032-01-01 (Estimated); Study Completion 2032-01-01 (Estimated)

PRIMARY OUTCOMES:
Collection of biological specimens to assess host microbiome response | Through End of Study
  To provide samples for use in secondary research for evaluation of assay validation, optimization of techniques for collection, storage, processing and analyzing samples, control samples for research tests in other studies, and identification of potential targets from which clinical trials can be designed to better understand or mitigate microbiome associated diseases

CONTACTS AND LOCATIONS:
Overall Officials: Suchitra K Hourigan, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001146-I.html